CLINICAL TRIAL: NCT06762236
Title: Combined Effects of Inspiratory Muscles Training With Pilate Training on Dyspnea Cardiorespiratory Fitness Quality of Life in Asthma Patients
Brief Title: Combined Effects of Inspiratory Muscles Training With Pilate Training in Asthma Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dureshawar Alamgir
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Asthma
Keywords: asthma patient, cardiorespiratory fitness, dyspnea, quality of life, Pilate training, inspiratory muscle training
MeSH Terms: conditions — Asthma; Dyspnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): .The session will repeated three times per week for 6 weeks with 40-minute sessions In Pilates we include 5 Pilate exercise, The Hundred (Rhythmic Breathing), Single Leg Stretch (Rhythmic Breathing), side kick, Toe Taps (Set Breathing Pattern) ,leg pull front for 6 weeks.
  Interventions: Other: Pillatate Training
- Controlied Group (Placebo Comparator): Inspiratory training, incentive spirometer the participants were instructed to hold the breath for 2-3 seconds then exhale slowly. This process was repeated 10 times or about 10-15minutes with rest in between 30 seconds. Base line treatment is diaphragmatic breathing exercise
  Interventions: Other: Pillatate Training

INTERVENTIONS:
Other: Pillatate Training — .The session will repeated three times per week for 6 weeks with 40-minute sessions In Pilates we include 5 Pilate exercise, The Hundred (Rhythmic Breathing), Single Leg Stretch (Rhythmic Breathing), side kick, Toe Taps (Set Breathing Pattern) ,leg pull front for 6 weeks.

SUMMARY:
Asthma is a chronic (long-term) condition that affects the airways in the lungs. The airways are tubes that carry air in and out of your lungs. In asthma the airways can become inflamed and narrowed at times. This makes it harder for air to flow out of your airways when you breathe out. When symptoms get worse, it is called an asthma attack. There is no permeant cure for asthma, but medical treatment and physiotherapy treatment can help to manage it. There is many physiotherapy protocols can be used for asthma patients like aerobic exercises, breathing exercise etc. The objective of our study is determine the combine effects of inspiratory muscle training with Pilate training on dyspnea, cardiorespiratory fitness and quality of life in asthma patients.

The randomized control trial will used as study design as study design for this this purpose simple random sampling technique will be used to allocate the sample in two group The sample size will be calculated by the G-power analysis. This study will conduct in Jinnah Hospital, Lahore Group A will receive both inspiratory training and Pilate training and group B receive only Inspiratory training, incentive spirometer the participants were instructed to hold the breath for 2-3 seconds then exhale slowly. This process was repeated 10 times or about 10-15minutes with rest in between 30 seconds. Base line treatment is diaphragmatic breathing exercise .The session will repeated three times per week for 6 weeks with 40-minute sessions In Pilates we include 5 Pilate exercise, The Hundred (Rhythmic Breathing), Single Leg Stretch (Rhythmic Breathing), side kick, Toe Taps (Set Breathing Pattern) ,leg pull front. Pre and post measurement will be done using Juniper asthma quality of life, 6 mint walk test, Borges dyspnea scale and fatigue severity scale to measure the outcomes. Data will be analyzed SPSS version 25. T-test and Regression analysis will be used.

Key words: asthma patient, cardiorespiratory fitness, dyspnea, quality of life, Pilate training, inspiratory muscle training

DETAILED DESCRIPTION:
To determine the combined effects of inspiratory muscles training with Pilate training on dyspnea, cardiorespiratory fitness quality of life in asthma patients

ELIGIBILITY:
Inclusion Criteria:

* Age range from 30 to 50 (15)
* Both Male and Female
* FEV1 value range from 64% to less than 50%
* Medically cleared for cardiac rehabilitation.
* Medical treatment, for at least 6 months
* Clinically stable (i.e., no exacerbation or medication changes for at least 30 days.

Exclusion criteria

* Status Asthmatics
* Patient with cardiac disease
* Age range from 30 to 50 (15)
* Both Male and Female
* FEV1 value range from 64% to less than 50%
* Medically cleared for cardiac rehabilitation.
* Medical treatment, for at least 6 months
* Clinically stable (i.e., no exacerbation or medication changes for at least 30 days.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
SF 36 | 8 weeks
  A disease-specific health-related quality of life instrument developed by E. Juniper in1999and colleagues that taps both physical and emotional impact of disease. The instrument should not be confused with the measure developed by Marks and colleagues, which carries the same name. Asthma Quality of Life Questionnaire (AQLQ or AQLQ-J) developed by Juniper and colleagues is a 32 questions instrument to measure the functional problems that are most troublesome to adults. Symptoms (11 items), Activity Limitation (12 items, 5 of which are individualized), Emotional Function (5 items), and Environmental Exposure (4 items) Scaling of items 7-point Likert scale Scoring All items are weighted equally. Mean score is calculated across all items within each domain. Overall score is the mean across all items
6MWT | 8 weeks
  The 6MWT is a sub-maximal exercise test used to examine person aerobic capacity and endurance. This test initially developed to make an assessment of patient with cardiopulmonary issues. It is used to check the functional capacity of the individual and it provides useful information regarding all the body systems during physical activity, including cardiovascular and pulmonary system. It can used for all age group range 2 to above 64 years The test is easy to perfume , with standardized limited instructions and encouragement being given as person walk as far as possible over 6 minutes through a flat corridor. The final distance is recorded in meters6

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Hameed, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No